CLINICAL TRIAL: NCT02490267
Title: Health- and Vision-Related Quality of Life in Children and Young People With Childhood Glaucoma, Childhood Cataract and Congenital Eye Defects
Brief Title: Quality of Life in Children Glaucoma and Cataract
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DALA1020
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Paediatrics With Cataracts; Paediatrics With Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: children with primary or secondary glaucoma
  Interventions: Other: Quality of Life questionnaire
- 2: children w/ cataract or previously treated for cataract
  Interventions: Other: Quality of Life questionnaire
- 3: children w/ microphthalmia, anophthalmia or coloboma
  Interventions: Other: Quality of Life questionnaire
- control group: age matched children without eye and vision problems.
  Interventions: Other: Quality of Life questionnaire

INTERVENTIONS:
Other: Quality of Life questionnaire

SUMMARY:
The management of childhood glaucoma (CG), childhood cataract (CC) and other birth defects affecting the eyes requires frequent hospital attendances and often multiple surgical and medical interventions, and are often associated with poor vision. Chronic medical conditions and vision impairment can affect quality of life (QoL). The QoL of children with the above conditions has not previously been evaluated.

DETAILED DESCRIPTION:
We wish to evaluate health related and vision related quality of life (HRQoL, VRQoL) in children age 2 to 16 years with childhood glaucoma (CG), childhood cataract (CC) and congenital eye defects microphthalmia, anophthalmia or coloboma (MAC).

We will recruit children who attend the children's eye clinics at Moorfields Eye Hospital at City Road. We will include the following subgroups:

A) children with primary or secondary glaucoma B) children with cataract or previously treated for cataract C) children with microphthalmia, anophthalmia or coloboma D) control group: agematched children without eye and vision problems. We will ask children and their carers to complete two age appropriate, validated questionnaires, the PedsQL (health related quality of life) and the Cardiff Visual Ability Questionnaire for Children. From the medical notes, we will record diagnosis and best corrected visual acuity with both eyes open. We will also record details of previous and current treatment, such as number of previous surgical interventions (sum of interventions right and left eye) and number of current topical medications (sum of eyedrop applications per day right and left eye).

ELIGIBILITY:
Inclusion Criteria:

A) children with primary or secondary glaucoma B) children with cataract or previously treated for cataract C) children with microphthalmia, anophthalmia or coloboma D) control group: age-matched children without eye and vision problems

Exclusion Criteria:

* Ocular hypertension not requiring treatment; visually not significant cataract; inability to communicate in English; surgical intervention (incisional) within one month of potential date of completing questionnaire (before or after)

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will recruit children who attend the children's eye clinics at Moorfields Eye Hospital at City Road. We will recruit children with healthy eyes and normal vision amongst the siblings who accompany new patients in Child Vision Clinics and the paediatric A&E. This approach will ensure that families have not previously been burdened with frequent hospital appointments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Incidence of babies requiring treatment for retinopathy of prematurity in the UK. | 1 year
  Captured in questionnaire

SECONDARY OUTCOMES:
Demographic characteristics of babies that need treatment, | 1 year
  Captured in questionnaire
Outcome of the treatment at 1 year follow up: anatomical and functional | 1 year
  Captured in questionnaire
Type of treatment administered | 1 year
  Captured in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, Dr Med PhD, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, London, United Kingdom